CLINICAL TRIAL: NCT04439396
Title: Use of Perioperative Ketorolac in Breast Surgery to Reduce Post Operative Pain and Opioid Use
Brief Title: Toradol (Ketorolac) in Breast Surgery to Reduce Pain & Opioid Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, James T Thompson, Plastic and Reconstructive Surgeon, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-387
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Breast Reduction; Breast Reconstruction
MeSH Terms: interventions — Ketorolac Tromethamine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: randomized
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Saline injection administered during surgical procedure
  Interventions: Other: Saline
- Low Dose (15mg) Toradol (Experimental): 15mg ketorolac (toradol) administered during surgery
  Interventions: Drug: Ketorolac Tromethamine
- High Dose (30mg) Toradol (Experimental): 30mg ketorolac (toradol) administered during surgery
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — nonsteroidal anti-inflammatory drug
  Other Names: Toradol
  Arms: High Dose (30mg) Toradol; Low Dose (15mg) Toradol
Other: Saline — saline fluid injection
  Arms: Control

SUMMARY:
The purpose of this study is to investigate whether perioperative single-dose administration of ketorolac (Toradol) can reduce post-operative pain after breast surgery, thereby decreasing post-operative opioid use.

DETAILED DESCRIPTION:
The investigators will perform a double blinded, prospective randomized trial of perioperative ketorolac (Toradol) on breast reduction and breast reconstruction procedures. Patients will be randomized into three groups: group 1 will receive a perioperative dose of ketorolac (Toradol, 15mg), group 2 will receive ketorolac (Toradol, 30mg), and group 3 will be the control and receive a placebo of saline. Patients will be asked to complete a diary or log of their average pain and pain medication use to be turned in at a 2 week follow up visit.

The patients, surgeons, anesthesiologist will not know whether the patient received ketorolac (Toradol) intraoperatively. Patients' pain will be assessed using pain scores in the immediate post-operative period, on post-operative day 1, and at their two-week follow up appointment. If patients leave the same day then they will only have two pain score assessments; on day of surgery and at their two-week follow up. Additionally, patients will be asked to assess their average pain (scale of 1-10 with 1 being no pain and 10 being extreme pain) in morning and evenings using a patient diary for the two week post-op period. The patient's opioid use will be measured by their opioid use during their hospital stay, as well as how many prescription narcotic pills the patient used to manage their pain at home, as documented using the patient diary.

ELIGIBILITY:
Inclusion Criteria:

* Patient consents to study
* Adult females needing breast reconstruction or breast reduction (day surgeries)

Exclusion Criteria:

* Patients with known kidney disease
* Patient does not consent
* patients with history of bleeding disorder, peptic ulcer disease, renal disease, blood thinners use, bariatric surgery and any other contraindications of Toradol use
* patients currently taking aspirin
* pregnant women (not standard to operate on this population anyway)

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Change of post-operative pain: Likert scale | 2 week post operation
  This will be assessed by using a Likert scale(0=no pain to 10=extreme pain) for pain in the post-operative period before they are discharged. If patients are kept overnight then another pain assessment will be done. Additionally, patients will keep a 2-week diary of average pain in the morning and evening each day until their 2 week follow up visit.

SECONDARY OUTCOMES:
Change of narcotic use | 2 weeks post operation
  This will be assessed by calculating the Medial Morphine Equivalent (MME) in the post-operative period. This will include narcotics given while in the hospital and narcotics prescribed and used at home in the patient diary. Perioperative narcotic use will also be recorded.
Complication assessment | 2 weeks to 90 days post operation
  Assess complications including, but not limited to, hematomas, GI issues (nausea, diarrhea, indigestion, heartburn), and headaches. This will be assessed by tracking any readmissions for hematoma evacuation or other complications reported at their post-op follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: James Thompson, Principal Investigator — Carilion Clinic
Locations (1):
- James T. Thompson, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No